CLINICAL TRIAL: NCT00184587
Title: Prophylactic Treatment of Episodic Cluster Headache With an Angiotensin II Receptor Blocker (Candesartan Cilexetil); a Randomized, Placebo Controlled Parallel Study
Brief Title: Prophylactic Treatment of Episodic Cluster Headache
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2452L0004; 2004-002737-39 (EudraCT Number); 045-04 (Other: Norwegian National Headache Centre); 10815 (Other: NSD)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2010-09

CONDITIONS: Cluster Headache
Keywords: prophylactic; episodic; cluster; candesartan; angiotensin II receptor blocker; randomized placebo controlled parallel study; headache diary
MeSH Terms: conditions — Cluster Headache; Recurrence | interventions — candesartan cilexetil; Angiotensin Receptor Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- candesartan (Experimental): candesartan cilexetil 16 mg (one tablet/day) in week 1 and 32 mg (2 tablets/day) in week 3, provided for the study by AstraZeneca
  Interventions: Drug: candesartan cilexetil
- placebo (Placebo Comparator): placebo one tablet/day in week 1 and 2 tablets/day in week 3, provided for the study by AstraZeneca. Same size, weight, taste and appearance as experimental drug
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: candesartan cilexetil
  Other Names: angiotensin II receptor blocker
  Arms: candesartan
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether candesartan cilexetil are effective prophylactic treatment of episodic Cluster headache

DETAILED DESCRIPTION:
Cluster headache is an unilateral headache with periodic attacks, that usually lasts for 6 to 12 weeks. The pain is usually unbearable. The attacks are treated with injections of sumatriptan (migraine medication)and inhalation of oxygen.

The most common prophylactics today has limited effect and a risk of side effects.

Candesartan has in one study shown a clinically significant effect in migraine prophylaxis.

The angiotensin II receptor blocker, candesartan is well tolerated with side-effects not significantly different from placebo and with few drug interactions. We therefore wish to investigate the prophylactic effect in treatment of cluster in headache patients.

This will be a multicenter, double-blind, randomized, parallel study where the prophylactic effect of candesartan is compared to placebo in a period of 3 weeks. First week 16 mg and the following 2 weeks 32 mg.

ELIGIBILITY:
Inclusion Criteria:

* The episodic cluster headache must be diagnosed according to the IHS classification. Had at least one episode with cluster headache before inclusion. Previously had at least one cluster headache episode lasting one month or more. At the time of inclusion, the cluster headache period shall not have lasted more than 3 weeks

Exclusion Criteria:

* Pregnancy, nursing, decreased hepatic og renal function, psychiatric illness, cardiac problems, hypersensitivity to candesartan, previous serious allergic reaction to medication, chronic cluster headache, drug/alcohol abuse, use of antipsychotic,antidepressants, lithium or other prophylactic treatment less than one month prior to inclusion, systolic blood pressure below 110 mmHg, use of other hypertensive medication, use og other specific attack medication than sumatriptan injection or oxygen 7-10l/min and inability to change medication, use of other triptans than sumatriptan during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-03; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
frequency of attacks per week | change from 'pseudobaseline' week 1 to week 3

SECONDARY OUTCOMES:
level of disability | change from 'pseudobaseline' week 1 to week 3
  5-point scale; 0= no disability, 1= mild, 2= moderate, 3= severe, 4= unbearable
duration of attacks | change from 'pseudobaseline' week 1 to week 3
hours with cluster headache | change from 'pseudobaseline' week 1 to week 3
days with cluster headache | change from 'pseudobaseline' week 1 to week 3
occurrence of autonomic symptoms | change from 'pseudobaseline' week 1 to week 3
number of treatments with sumatriptan or oxygen | change from 'pseudobaseline' week 1 to week 3
patient satisfaction with treatment | change from 'pseudobaseline' week 1 to week 3
  scale from 1 to 10 with 1= very poor effect and 10= very good effect
headache severity index | change from baseline to 1 week and 3 week
  product of level of disability and duration of attacks
candesartan-responders | 3 weeks
  patients with a 50% or more reduction in attack frequency in week 3 than in week 1
placebo-responders | 3 weeks
  patients with a 50% or more reduction in attack frequency in week 3 than in week 1

CONTACTS AND LOCATIONS:
Overall Officials: Lars J Stovner, PhD, Principal Investigator — Norwegian National Headache Center St.Olavs Hospital
Locations (1):
- Norwegian National Headache Centre St.Olavs Hospital, Trondheim, Trondheim, Norway

REFERENCES:
- [Background] Tronvik E, Stovner LJ, Helde G, Sand T, Bovim G. Prophylactic treatment of migraine with an angiotensin II receptor blocker: a randomized controlled trial. JAMA. 2003 Jan 1;289(1):65-9. doi: 10.1001/jama.289.1.65. PMID 12503978
- [Result] Tronvik E, Wienecke T, Monstad I, Dahlof C, Boe MG, Tjensvoll AB, Salvesen R, Zwart JA, Jansson SO, Stovner LJ. Randomised trial on episodic cluster headache with an angiotensin II receptor blocker. Cephalalgia. 2013 Sep;33(12):1026-34. doi: 10.1177/0333102413484989. Epub 2013 Apr 18. PMID 23598371